CLINICAL TRIAL: NCT04478435
Title: The Comparative Gastric Volume Estimation Between Different Time Intervals by Ultrasonography After Glucose Loaded Clear Fluid Ingestion in Fasted Healthy Adult
Brief Title: Gastric Volume Estimation by Ultrasonography After Glucose Loaded Clear Fluid Ingestion in Fasted Adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FF-2018-447
Record Dates: First submitted 2020-07-05; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Healthy Participants
Keywords: gastric antrum ultrasonography; Gastric volume estimation; aspiration risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 Hour post intervention (Active Comparator): Ultrasound assessment done 1 hour after ingestion of glucose loaded drink
  Interventions: Other: glucose loaded clear fluid
- 2 hours post intervention (Placebo Comparator): Ultrasound assessment done 2 hour after ingestion of glucose loaded drink
  Interventions: Other: glucose loaded clear fluid

INTERVENTIONS:
Other: glucose loaded clear fluid — Ultrasound assessment of gastric antrum is done at different time interval following glucose loaded clear fluid ingestion

SUMMARY:
Introduction; Pre operative gastric ultrasonography is a newly developed tool used to evaluate gastric content and volume in assessing perioperative aspiration risk and guide anaesthetic management. Gastric antrum is the most amenable and most consistently identified region for sonographic examination during assessment even in empty state. Baseline gastric secretions and clear fluids i.e: water, apple juice and tea have hypoechoeic or anechoic appearance, whilst milk, thick fluids, or suspensions will have increased echogenicity. Evaluation with sonographic assessment were found to be accurately reflective of gastric content in various studies.

In this study, healthy volunteers were recruited. They will be required to fast at least 8 hours prior to baseline gastric antrum ultrasonography assessment. Following that, they will require to drink 250ml glucose loaded drinks. Repeated Ultrasound assessment will be done after 1 hour of glucose loaded drink ingestion in Group 1 and after 2 hours in Group 2. Hypothesis of the study is there will be no significant different between ultrasound assessment between this 2 groups.

DETAILED DESCRIPTION:
This prospective randomized controlled trial study will be conducted in the Department of Anaesthesiology and Intensive Care UKM for eight months period from November 2018 to June 2019 involving healthy adult volunteers comprising staff members of Department of Anaesthesiology and Intensive Care, after obtaining approval from Research Committee of the Department of Anaesthesiology & Intensive Care, Hospital Canselor Tuanku Muhriz, Universiti Kebangsaan Malaysia Medical Centre (UKMMC) and the Medical Research & Ethics Committee, UKMMC. Written informed consent will be obtained from volunteers who fulfill the inclusion criteria.

All volunteers will be fasted, a minimum of 8 hours (duration of fasting will be recorded before the study begin) and will undergo baseline ultrasonographic gastric assessment (t0).

All subjects in Group 1 and group 2 will drink 250 ml of lychee juice (glucose loaded clear fluid containing solution with lychee flavor; 145 kcal in 250 ml) after completion of baseline gastric assessment.

Group 1 subjects will then continue fasting for one hour until completion of second sonographic antral assessment. Subjects in Group 2 will continue fasting for 2 hours until second sonographic antral assessment scan is completed.

Subjects will be divided into 2 groups via computer randomization which will be allocated by anaesthesia trainee that will not be taking part in the analytical and further write up phases of the study. Ultrasonographic volume assessment will be conducted by a single operator who is an anaesthesia Masters trainee, experienced in diagnostic abdominal ultrasound with more than 20 sonographic gastric volume assessments. The images will be recorded and validated by a consultant radiologist.

Ultrasonographic views of antral area will be obtained using a curvilinear array 2- to 5-MHz transducer and a Mindray DC-70 (Shanghai, China) with image compounding technologies. Images will be obtained with the stomach at rest, and between peristaltic contractions. Sonograms of the antral area will be examined in 2 views, cross-section in the supine position, followed by the right lateral decubitus position, at each of the two scanning sessions.

During ultrasonography, the antrum will be imaged in a parasagittal plane in the epigastric area using the left lobe of the liver, the inferior vena cava, and the superior mesenteric vein as internal landmarks. The two vessels are usually visualized slightly to the right of the abdominal midline. Once these vessels were identified, the transducer will be rotated slightly clockwise or counterclockwise to best obtain a true cross-sectional view of the antrum. The anteroposterior and craniocaudal diameters will be measured in this view.

CSA of the antral area (a two-dimensional section) will be calculated according to the formula previously used by Bolondi18 using two maximum perpendicular diameters.

This formula essentially represents the surface area of an ellipse, as follows: CSA (AP x CC x pie/4), where AP is the anteroposterior diameter and CC is the craniocaudal diameter measures in one decimal point.

Estimation of gastric volume will be obtain using this formula:

Predicted gastric volume based on right lateral CSA value : 27 + 14.6 * right lat CSA - 1.28*age (negative volume value indicates and empty state).

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 & 2

Exclusion Criteria:

* Upper gastrointestinal pathology such as hiatus hernia, oesophageal cancer
* Prior surgery to upper GI
* On medication that may affect gastric emptying time
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 254 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Gastric volume assessment | 1 hour after intervention
  Gastric volume can be calculated with gastric antrum measurement
Gastric volume assessment | 2 hours after intervention
  Gastric volume can be calculated with gastric antrum measurement

OTHER OUTCOMES:
Baseline gastric volume | Baseline
  Baseline gastric volume assessed prior to ingestion of glucose loaded clear fluid

CONTACTS AND LOCATIONS:
Overall Officials: Syarifah Noor Nazihah S Masri, Principal Investigator — PPUKM
Locations (1):
- Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur, Wp, Malaysia

IPD SHARING:
Plan to Share IPD: No
IPD will be share on request

REFERENCES:
- [Result] Warner MA, Warner ME, Weber JG. Clinical significance of pulmonary aspiration during the perioperative period. Anesthesiology. 1993 Jan;78(1):56-62. doi: 10.1097/00000542-199301000-00010. PMID 8424572
- [Result] Read MS, Vaughan RS. Allowing pre-operative patients to drink: effects on patients' safety and comfort of unlimited oral water until 2 hours before anaesthesia. Acta Anaesthesiol Scand. 1991 Oct;35(7):591-5. doi: 10.1111/j.1399-6576.1991.tb03354.x. PMID 1785235
- [Result] Perlas A, Davis L, Khan M, Mitsakakis N, Chan VW. Gastric sonography in the fasted surgical patient: a prospective descriptive study. Anesth Analg. 2011 Jul;113(1):93-7. doi: 10.1213/ANE.0b013e31821b98c0. Epub 2011 May 19. PMID 21596885
- [Result] Kruisselbrink R, Gharapetian A, Chaparro LE, Ami N, Richler D, Chan VWS, Perlas A. Diagnostic Accuracy of Point-of-Care Gastric Ultrasound. Anesth Analg. 2019 Jan;128(1):89-95. doi: 10.1213/ANE.0000000000003372. PMID 29624530